CLINICAL TRIAL: NCT03258606
Title: Characteristics and Outcomes of a Capacity-to-Consent Assessment Service
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 999917119; 17-CC-N119
Record Dates: First submitted 2017-08-22; First posted 2017-08-23 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Dysfunction
Keywords: Surrogate; Decision Making; Capacity to Consent; Cognitive Impairment; Enrollment; Natural History
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Individuals with affected capacity to consent: Individuals with who were unable to consent and were allowed by protocol to give surrogate consent.

SUMMARY:
Background:

Many medical conditions such as Alzheimer s disease limit the ability of people to think clearly. For medical scientists to best study these medical conditions, they need to enroll some people who may not be able to consent to participate in research on their own. Before these individuals enroll in research it is important to assess whether they are able to consent or whether someone else will need to consent for them. The NIH Clinical Center has a team that performs these assessments. A team like this can be useful for two reasons. First, it helps to protect the rights of research participants. Second, it makes it possible to study medical conditions that could not be studied otherwise. In this study we will look back at the records of the NIH Clinical Center team to review the process and results of these assessments. We expect to learn how the capacity assessments were done. We will learn what factors make people more or less able to consent. We will learn who consented for the research participants when they could not consent on their own, for example a spouse or an adult child. These results are likely to be useful to other researchers who wish to study diseases that limit cognitive ability.

Objective:

To study the process and outcomes of capacity assessments of people who may not be able to consent to research.

Eligibility:

People of all ages, genders, races, ethnicities, and languages whose ability to consent was assessed at the NIH Clinical Center at some time during the years 1999-2016.

Design:

This study will only review existing records. There will not be any active participants.

Records will be reviewed for research only. This will take place in the Clinical Center. It will be done by staff of the Department of Bioethics and the Human Subjects Protection Unit (HSPU).

The study will collect data from the Bioethics Consult database. It will also collect data from HSPU records.

Researchers will look at demographic data. They will look at details of capacity evaluations.

Personal data will not be extracted from existing records.

DETAILED DESCRIPTION:
Objective: To characterize the process and outcomes of capacity assessments of individuals who may be unable to consent to participate in research.

Study population: all individuals who came to the NIH Clinical Center for possible enrollment in research whose capacity to consent or assent was evaluated by the Bioethics Consultation Service (BCS), the Human Subjects Protection Unit (HSPU), or the Ability to Consent Assessment Team (ACAT), and all surrogate decision makers of individuals who were unable to consent and were allowed by protocol to give surrogate consent.

Design: Retrospective record review

Outcome measures: The primary outcome measure will be whether prospective research participants were judged to be able to consent or not. Secondary measures will include: whether the consulting team considered it ethically acceptable to enroll the participant in research; how consent was obtained for doing so; and descriptive features of the consults such as the Institute that requested the consult, protocols for which consults were requested, and diseases that prompted capacity assessments, among other descriptive characteristics.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant ages 7 to 99
* Participants must have undergone some type of capacity evaluation, consent or assent monitoring, or surrogate assessment, by the BCS, HSPU, or ACAT.
* Children (or adults) who were seen by the consultation service for the purposes of either evaluating their ability to assent or for assent monitoring

Exclusion Criteria:

-Pregnant women or prisoners will not be included

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals who came to the NIH Clinical Center for possible enrollment in research whose capacity to consent or assent was evaluated by the Bioethics Consultation Service (BCS), the Human Subjects Protection Unit (HSPU), or the Ability to Consent Assessment Team (ACAT), and all surrogate decision makers of individuals who were unable to consent and were allowed by protocol to give surrogate consent.
Sampling Method: Non-Probability Sample
Enrollment: 1098 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Whether prospective research participants were judged to be able toconsent or not. | At record review
  Whether the consulting team considered it ethically acceptable to enroll the participant in research and how consent was obtained for doing so.

SECONDARY OUTCOMES:
Other measures that will be collected include demographics, results of the evaluation, kinds of research conducted and content of capacity assessments. | At record review
  Other measures that will be collected include demographics, results of the evaluation, kinds of research conducted and content of capacity assessments.
Whether the consulting team considered it ethically acceptable toenroll the participant in research and how consent was obtained for doing so. | At record review
  Whether the consulting team considered it ethically acceptable to enroll the participant in research and how consent was obtained fordoing so.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Danis, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States